CLINICAL TRIAL: NCT06535178
Title: Determining the Influence of Sleep on Cardiovascular Outcomes
Brief Title: The Influence of Sleep on Cardiovascular Outcomes
Acronym: DISCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medical Research Foundation, Oregon (Other)
Responsible Party: Principal Investigator, Andrew McHill, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00026854
Record Dates: First submitted 2024-07-31; First posted 2024-08-02 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Circadian Rhythm; Cardiometabolic Health; Vascular Health; Pain
Keywords: Circadian Rhythm; Cardiometabolic Health; Vascular Health; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Regularity Group (Experimental): Individuals in the lowest SRI tertile will begin the 12-week intervention to improve sleep regularity. Participants will be instructed to maintain a consistent sleep onset time (±30 min self-selected sleep time).
  Interventions: Behavioral: Sleep Regularity Group
- Control Group (No Intervention): All other participants will be instructed to maintain their habitual sleep patterns.

INTERVENTIONS:
Behavioral: Sleep Regularity Group — Maintained consistent sleep onset time (±30 min self-selected sleep time) for 12-weeks.
  Arms: Sleep Regularity Group

SUMMARY:
The goal of this study is to identify the effects of sleep regularity on cardiovascular regulatory mechanisms. The investigators are hoping to discover if improving the regularity of sleep timing will improve metabolic and vascular health markers. The protocol is a 12-week prospective cohort study that includes both field and in-laboratory data collection in ostensibly healthy male and female adults, aged 18-40years. We will also have a sub-group of individuals with chronic pain to examine the effects of sleep regularity on pain outcomes.

DETAILED DESCRIPTION:
Sleep is a fundamental determinant of heath; however, the impact of day-to-day variations in sleep patterns (i.e., sleep regularity) on cardiometabolic and vascular health has been underappreciated. Emerging evidence suggests that less regularity in sleep timing is correlated with cardiometabolic health and is a stronger predictor of mortality risk than sleep duration. In this cohort, the investigators will determine the influence of sleep regularity on mechanisms that impact cardiometabolic, vascular, and autonomic function.

The misalignment of behaviors (e.g., sleep) with the internal timing system (i.e., circadian misalignment) is likely a mechanistic contributor to unfavorable health outcomes. Laboratory experiments have shown that acute circadian misalignment increases markers of inflammation, alters metabolism, and elevates mean arterial pressure. We have shown that poorer overnight blood pressure dipping patterns are associated with circadian disruptions elicited by decreased sleep regularity, which occurs within 90-days of transitioning to a shift work schedule. There is a need to characterize the influence of sleep regularity on the underlying pathways that affect health.

The goal of this study is to determine the effect of an intervention targeting improved sleep regularity on circadian, metabolic, and vascular health markers. Participants within the lowest tertile for sleep regularity will adhere to a consistent sleep onset time (±30 min) for approximately 12-weeks. The outcomes that the investigators will focus on will be indices of hemodynamics (blood pressure, heart rate, autonomic function), blood biomarkers (markers of inflammation, oxidative stress, and triglycerides), energy metabolism, weight, and percent body fat. We will also have a sub-group of individuals with chronic pain to examine the effects of sleep regularity on pain outcomes.

1. Outpatient Biobehavioral Weeks: Actigraphy data will be collected across 2-weeks to assess habitual sleep patterns and calculate a sleep regularity index (SRI).
2. Biobehavioral Laboratory Visit: Participants will be asked to visit the OHSU School of Nursing (SON) Biobehavioral Laboratory space for two in-laboratory visits in dim-light settings, which will involve an evening stay (~7.5h) to measure circadian markers, body composition, vascular function, and questionnaire data. Saliva samples will also be collected via salivettes in order to measure the hormone melatonin and determine each participants' dim-light melatonin onset (DLMO). Participants lowest SRI tertile (intervention group) will be instructed to maintain a consistent sleep onset time (±30 min self-selected sleep time) for up to 12-weeks. Compliance will be assessed across 6-weeks of outpatient bio-behavioral data collection via sleep logs, actigraphy, and daily surveys (described below). All other participants (control group) will be instructed to maintain their habitual sleep patterns for up to 12-weeks.
3. Ambulatory Monitoring: For participants in the intervention group, biobehavioral data collection will occur at Weeks 1-2, Weeks 6-7, and Weeks 11-12. For the control group, biobehavioral data collection will occur at Weeks 11-12. During these weeks, participants will wear an actigraphy device and keep sleep logs for 2-weeks during the biobehavioral data collection. Participants will also wear an ambulatory blood pressure cuff. Additionally, to measure glucose levels throughout the protocol, participants will be fitted with a continuous glucose monitor. Participants will complete daily surveys each bio-behavioral period to measure self-reported bed and wake times and naps.
4. Blood Biomarkers: At baseline and at Week 12, participants will visit the SON Biobehavioral Laboratory for a blood draw to obtain markers of inflammation, oxidative stress, and lipemic markers that will be measured with an ~10mL blood draw.

ELIGIBILITY:
Inclusion Criteria:

* Ostensibly healthy men and women Subgroup study (chronic pain)
* Satisfies diagnostic criteria for fibromyalgia according to the Widespread Pain Index - Symptom Severity (WPI-SS) scale with the following three conditions being met:

  1. Widespread pain index (WPI) ≥7 and symptom severity (SS) scale score ≥5 or WPI 3-6 and SS scale score ≥9.
  2. Symptoms have been present at a similar level for at least 3 months.
  3. The patient does not have a disorder that would otherwise explain the pain.

Exclusion Criteria:

* No history of drug or alcohol dependency.
* Must be current non-smokers, and are required to have a history of less than 5 pack years of smoking.
* No history of working irregular day and night hours, regular night work, or rotating shift work for the 1 year prior to the study. In addition to this, individuals must not have traveled across more than 1 time zone during the 3 months prior to the study.
* Chronobiologic and sleep disorders.
* Diseases of the cardiovascular system.
* Hypertension. Individuals will be allowed to be normotensive (resting systolic blood pressure of <140/90 mmHg, measured on more than one occasion) or uncomplicated stage 1 hypertension (systolic BP between 140 and 159 mmHg or a diastolic BP between 90 and 99 mmHg).
* Disorders of the respiratory system.
* Pre-diabetes/Diabetes. For participants who have self-reported pre-diabetes/diabetes.
* Disorders of the kidney and urinary tract.
* Infectious diseases.
* Disorders of the gastrointestinal system.
* Disorders of the immune system.
* Disorders of the hematopoietic system.
* Neoplastic diseases.
* Endocrine and metabolic diseases.
* Neurologic disorders.
* Must not be participating in another research study that would influence their safe participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in dim-light melatonin onset | Week 0 and Week 12
  Saliva samples will be collected pre- and post-12-week intervention and will be assayed for melatonin using standardized assays. Dim-light melatonin onset will be calculated using the linear interpolated point in time in which each participant's melatonin crosses and remains elevated above a 4pg/mL threshold. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in SRI | Week 0 and Week 12
  SRI will be calculated from 2-weeks actigraphy data prior to the first in-laboratory visit. Changes in SRI will be measured for 2-weeks during Weeks 1-2, Weeks 6-7, and Weeks 11-12 for the intervention group and during Weeks 11-12 for the control group. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in vascular endothelial function | Week 0 and Week 12
  Vascular endothelial function will be assessed via flow mediated dilation pre- and post-12-week intervention. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in heart rate | Week 0 and Week 12
  Heart rate will be measured every ~30 minutes via a blood pressure cuff. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in blood pressure | Week 0 and Week 12
  Changes in resting blood pressure will be measured every ~30 minutes via ambulatory blood pressure machines for up to 48-hours during Weeks 1-2, Weeks 6-7, and Weeks 11-12 for the intervention group and Weeks 11-12 for the control group. Blood pressure patterns during the day and night will be assessed, as well as a contrast of day and nighttime blood pressure levels. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in resting cardiac vagal tone | Week 0 and Week 12
  High frequency power of the heart rate variability power spectrum will be used to estimate cardiac parasympathetic activity (vagal tone). These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in heart rate response to exercise | Week 0 and Week 12
  Beat by beat heart rate will be recorded during a Monark bicycle ergometer exercise test where workload will be increased every 3-min until ~75% age predicted heart rate max is achieved. Heart rate will be averaged at rest, during each 3-min stage, and each minute during a 2-minute recovery. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in blood pressure response to exercise | Week 0 and Week 12
  Beat by beat blood pressure will be recorded during a Monark bicycle ergometer exercise test. Blood pressure will be averaged at rest, during each 3-min stage, and each minute during a 2-minute recovery. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in energy metabolism | Week 0 and Week 12
  Resting energy expenditure and macronutrient oxidation will be measured via indirect calorimetry. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in glucose | Week 0 and Week 12
  Changes in glucose will be measures during Weeks 1-2, Weeks 6-7, and Weeks 11-12 for the intervention group and Weeks 11-12 for the control group. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.

SECONDARY OUTCOMES:
Changes in MDA | Week 0 and Week 12
  Changes in malondialdehyde [MDA] will be measured pre- and post-12-week intervention. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in TAC | Week 0 and Week 12
  Changes in total antioxidant capacity [TAC] will be measured pre- and post-12-week intervention. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in CRP | Week 0 and Week 12
  Changes in C-reactive protein [CRP] will be measured pre- and post-12-week intervention. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in triglycerides | Week 0 and Week 12
  Changes in triglycerides will be measured pre- and post-12-week intervention. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in percent body fat | Week 0 and Week 12
  Percent body fat will be assessed via dual x-ray absorptiometry [DEXA] and a Tanita body composition scale in all participants at baseline. Changes in percent body fat will be assessed via DEXA (Intervention Group) and Tanita body composition scale (Control Group) post-12-weeks. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in weight | Week 0 and Week 12
  Weight will be assessed via dual x-ray absorptiometry [DEXA] and a Tanita body composition scale in all participants at baseline. Changes in weight will be assessed via DEXA (Intervention Group) and Tanita body composition scale (Control Group) post-12-weeks. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in BMI | Week 0 and Week 12
  Body mass index [BMI] will be assessed via dual x-ray absorptiometry [DEXA] and a Tanita body composition scale in all participants at baseline. Changes in BMI will be assessed via DEXA (Intervention Group) and Tanita body composition scale (Control Group) post-12-weeks. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Changes in PIPR | Week 0 and Week 12
  Changes in post illumination pupil response [PIPR] will be measured using a near-infrared illumination and solid-state video pre-and post-12-week intervention. These data will be used to calculate mean differences and standard deviations between the control and intervention group for future experiments. Examined using planned comparison dependent t-tests to compare the changes pre- and post-12-weeks.
Subjective Pain | Week 0 and Week 12
  Participants will rate feelings of subjective pain on visual analog scales.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W McHill, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No